CLINICAL TRIAL: NCT02266056
Title: The Benefits of Deep Neuromuscular Block and Sugammadex in Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2014-0559
Record Dates: First submitted 2014-08-26; First posted 2014-10-16 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer
Keywords: deep neuromuscular block; sugammadex; laparoscopic colorectal surgery; hemodynamic change
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep neuromuscular relaxation (Experimental)
  Interventions: Drug: Deep neuromuscular block using rocuronium and reversal with suggamadex
- Moderate neuromuscular relaxation (Active Comparator)
  Interventions: Drug: Moderate neuromuscular block using rocuronium and reversal with suggamadex

INTERVENTIONS:
Drug: Deep neuromuscular block using rocuronium and reversal with suggamadex — Deep neuromuscular block and moderate neuromuscular block with Esmerone and reversal with bridion
  Arms: Deep neuromuscular relaxation
Drug: Moderate neuromuscular block using rocuronium and reversal with suggamadex — Moderate neuromuscular block and moderate neuromuscular block with Esmerone and reversal with bridion
  Arms: Moderate neuromuscular relaxation

SUMMARY:
Pneumoperitoneum, the use of carbon dioxide, presents some disadvantages, including a risk of hypercarbia and respiratory acidosis during surgery in the respiratory system, and of an increased mean arterial pressure and systemic vascular resistance due to sympathetic excitation in the cardiovascular system. 10~15 mmHg intra-abdominal pressure is required in order to achieve a pneumoperitoneum, and increased abdominal pressure following a pneumoperitoneum causes hemodynamic changes leading to a reduced cardiac function by increasing the left ventricular end systolic wall stress and the right and left ventricular filling pressure, while decreasing the stroke volume and cardiac index. The author compared the intra-abdominal pressure necessary to achieve a pneumoperitoneum under deep muscle relaxation and medium muscle relaxation in ten patients undergoing laparoscopic surgery for colorectal cancer as part of preliminary research. The results showed that deep muscle relaxation, compared to medium muscle relaxation, was able to lower the intra-abdominal pressure by an average of 5.6 mmHg (13.2 ± 0.8 vs 7.6 ± 1.1) and the inspiratory pressure by an average of 8. Above all, even after lowering the intra-abdominal pressure with deep muscle relaxation, the surgeon was able to maintain a view almost identical to the one afforded by medium muscle relaxation. However, up until now, no reports have clearly indicated the change in pneumoperitoneum pressure, the patient's hemodynamic change, post-operative recovery, and surgical prognosis depending on the depth of muscle relaxation.Against this background, this study aims to identify the degree to which intra-abdominal pressure in laparoscopic colorectal surgery can be reduced by deep muscle relaxation, and the corresponding advantages this method presents in terms of physiological changes such as hemodynamic and respiratory system changes. In addition, the study intends to examine the difference between deep muscle relaxation and medium muscle relaxation in terms of surgical prognosis, including their effects on post-operative pain and on the patient's recovery of intestinal mobility.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 80 scheduled to undergo laparoscopic colorectal or rectal surgery below the ASA class 3

Exclusion Criteria:

* Patients with neuromuscular disease/patients with a personal history or family history of malignant hyperthermia/patients with a serious heart, kidney (GFR < 60) or liver condition (ALT/AST > 100)/ patients who have had colorectal or rectal surgery/obese patients (BMI ≥35)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
intra-abdominal pressure | 5 minuits after pneumoperitoneum
  The difference of intra-abdominal pressure during peumoperitoneum between deep neuromuscular block and moderate neuromuscular block to identify the degree to which deep muscle relaxation can reduce intra-abdominal pressure while maintaining the surgeon's view in a laparoscopic colorectal surgery or laparoscopic rectal surgery, as well as examine the simultaneous hemodynamic changes and changes in the respiratory system.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University, College of Medicine, Yonsei Health System, Yonsei Cancer Center, Seoul, Seoul, South Korea